CLINICAL TRIAL: NCT06767319
Title: Comparison of Depth of Focus Testing Methods
Brief Title: Prospective, Multi-center, Non-interventional, Open Label, Randomized (Depth of Focus Testing Sequences), Clinical Study
Acronym: Sierra
Status: Completed | Type: Observational
Sponsor: Johnson & Johnson Surgical Vision, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: MDEV110SDVA
Record Dates: First submitted 2024-12-17; First posted 2025-01-09 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Depth of Focus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Testing Order: The difference in diopters of depth of focus range achieving a threshold of 0.20 logMAR between Trial lens vs. Chart testing method per pre-study IOL group.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — The difference in diopters of depth of focus range achieving a threshold of 0.20 logMAR between Trial lens vs. Chart testing method per pre-study IOL group.

SUMMARY:
The purpose of this clinical study is to evaluate the difference in depth of focus measured with two methods in patients implanted with either TECNIS 1-piece Monofocal IOL or TECNIS Eyhance IOL:

1. Trial lens method
2. Chart testing at appropriate focal distances (or viewing distances)

ELIGIBILITY:
Study Eye Inclusion Criteria:

1. Patients unilaterally or bilaterally implanted with a TECNIS non-toric/toric monofocal or TECNIS non-toric/toric Eyhance IOL;
2. Signed informed consent and HIPAA authorization or equivalent documentation necessary to comply with applicable privacy laws in U.S.;
3. Availability, willingness, and sufficient cognitive awareness to comply with examination procedures.
4. Adults (Minimum 22 years of age or older at the time of participation in the study);

Study Eye Exclusion Criteria

1. Patients within 30 days postoperative from surgery;
2. BCDVA worse than 20/32;
3. Posterior capsular opacification or other medical findings affecting best-corrected distance visual acuity (BCDVA) in the opinion of the investigator;
4. Clinically significant ocular surface disease that would affect study measurements based on investigator medical opinion;
5. Prior corneal refractive surgery (SMILE, LASIK, LASEK, RK, PRK, etc.);
6. Known ocular disease or pathology that, in the opinion of the investigator may affect visual acuity (macular degeneration, cystoid macular edema, diabetic retinopathy, glaucoma, retinal detachment etc.);
7. Be an employee (e.g., Investigator, Coordinator, Technician) or immediate family member of an employee (including partner, child, parent, grandparent, grandchild or sibling of the employee or their spouse) of the clinical site.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: As only one eye per subject will be enrolled in the study based on the eligibility criteria, up to 115 subjects will be enrolled to obtain data on approximately 80 subjects to account for approximately 30% screen failure rate.
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2024-12-18 (Actual); Primary Completion 2025-03-11 (Actual); Study Completion 2025-03-11 (Actual)

PRIMARY OUTCOMES:
The difference in diopters of depth of focus range achieving a threshold of 0.20 logMAR between Trial lens vs. Chart testing method per pre-study IOL group. | One day Visit study
  The difference in diopters of depth of focus range achieving a threshold of 0.20 logMAR between Trial lens vs. Chart testing method per pre-study IOL group.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Empire Eye & Laser Center, Bakersfield, California
  - Jones Eye Center, Sioux City, Iowa
  - Cleveland Eye Clinic, Brecksville, Ohio
  - Parkhurst NuVision, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Devices Companies have an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA project site at http://yoda.yale.edu
URL: http://yoda.yale.edu